CLINICAL TRIAL: NCT06584877
Title: Investigating How Childhood Tumours and Congenital Disease Develop
Status: Enrolling by invitation | Type: Observational
Sponsor: The Wellcome Sanger Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 207523
Record Dates: First submitted 2024-07-04; First posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-07

CONDITIONS: Childhood Tumor; Congenital Disorders
MeSH Terms: conditions — Neoplasms; Congenital, Hereditary, and Neonatal Diseases and Abnormalities | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Surplus tumour/tissue, adjacent normal tissue and bone marrow. New or stored blood or saliva samples. Semen (from adult males).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Research participant with tumour or congenital condition: The participant identified to have a tumour or congenital condition (a condition from birth) that is likely to be due to errors of the genetic code (DNA).
  Interventions: Other: sample collection; Other: Seeking consent and assent
- Relatives: parents, siblings or close relatives of the participant with the tumour or congenital condition.
  Interventions: Other: sample collection; Other: Seeking consent and assent

INTERVENTIONS:
Other: sample collection — Surplus material from surgery. New or stored blood or saliva. Semen (from adult males).
Other: Seeking consent and assent — Consent or assent from all participants to be included in the study. Consent from parent / guardian for inclusion of children in study (as primary participant or relative/sibling, as applicable).

SUMMARY:
Every cell and every organ in the human body derives from a fertilised egg. As the fertilised egg divides, a human being develops and grows. The process of how the fertilised egg divides and forms a human being is very sophisticated and is directed by the genetic information, the DNA, that is present in every cell.

When errors, mutations, in the DNA code arise, the orderly process of human development can be disrupted. This can lead to the development of tumours during childhood and congenital diseases (that is, abnormalities that children are born with).

The aim of this study is to define exactly which DNA errors underpin childhood tumours and congenital diseases.

DETAILED DESCRIPTION:
Cancers and some congenital anomalies are caused by changes (mutations) in the genetic code (DNA) of cells. The use of Next Generation Sequencing (NGS) has enabled the study of the genetic changes that underpin these diseases, genome wide and at base pair resolution.

A key question about the molecular pathogenesis of a range of childhood tumours and congenital anomalies that remains unanswered is the order in which the different mutations arise. To define the order in which mutations arise, the investigators will need to reconstruct the life history of individual tumours / anomalies. This can be achieved by segregating the major clone ('ancestral' cell) from sub-clones or by studying multiple areas from the same lesion. Although this approach allows timing of mutations to some degree, in childhood tumours and congenital lesions this approach is fundamentally limited by the inability to define embryonic mutations. The basis of the limitation is that the lesions in question is conventionally compared to the patient's germline (the genetic information they have from birth). In such a comparison embryonic mutations will be misclassified as either germline or somatic (acquired).

To overcome this limitation one would have to compare the lesion to the parental germline.

Thus, here this study proposes to perform the first NGS study of childhood tumours and congenital anomalies, focusing on defining the embryonic pathogenesis. A unique feature of this study will be that lesions will be compared to the parental germline to define embryonic mutations. A focus of the analysis will be to define order in which mutations arise.

ELIGIBILITY:
Inclusion Criteria:

* Presence of childhood tumour / congenital disease, or relative of participant with childhood tumour / congenital disease
* Sufficient 'surplus to diagnostic/clinical use' tissue is available
* Child assent and parental/guardian consent obtained where applicable

Exclusion Criteria:

* Insufficient surplus tissue is available

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will have either a tumour or congenital anomaly. The investigators aim to also recruit the participant's biological parents. In some cases, the participant's sibling(s) and close relatives may also be recruited into the study. Where post-mortem material will be accessed, the participant will have been enrolled in the study whilst alive.
  Potential participants will be identified by participating NHS clinicians on an ongoing basis and from registers of patients internal to each participating NHS unit.
  Surplus samples will be identified by participating NHS clinicians. Some samples may also be obtained through Biobanks.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-02-02 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Description of the genetic mutations of each tumour and congenital anomaly. | 9.5 years
  For each tumour a catalogue of mutations will be derived from sequencing reads. The catalogues will be compared across tumour types / anomalies to identify the mutations that drive individual tumour types / anomalies. The life history of each tumour / anomaly will be determined.
  Methylation data will be analysed to derive a methylation profile for each tumour. The profiles of individual tumours will then be compared with each other to see whether tumour-type specific methylation profiles exist.

CONTACTS AND LOCATIONS:
Overall Officials: Sam Behjati, PhD, Principal Investigator — The Wellcome Sanger Institute
Locations (1):
- Wellcome Sanger Institute, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No
As is customary in the field, we will publish our anonymised data in research databases and archives. This includes EGA (European Genome-phenome Archive) where data will be made accessible via managed access to researchers or companies worldwide.